CLINICAL TRIAL: NCT01702727
Title: Evaluation and Development of a Novel Binocular Treatment (I-BiTTM) System Using Video Clips and Interactive Games to Improve Vision in Children With Amblyopia ('Lazy Eye').
Brief Title: I-BiT - Evaluation of a Novel Binocular Treatment System (I-BiTTM) in Children With Amblyopia
Acronym: I-BiT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10OY006
Record Dates: First submitted 2012-08-08; First posted 2012-10-08 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Amblyopia
Keywords: Amblyopia; I-BiT TM; Interactive games; Binocular
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- I-BiTTM game (Experimental): 30 minutes intervention weekly for 6 weeks.
  Interventions: Device: I-BiTTM game
- Non-I-BiTTM game (Active Comparator): 30 minutes intervention weekly for 6 weeks.
  Interventions: Device: Non-I-BiTTM game
- I-BiTTM DVD (Experimental): 30 minutes intervention weekly for 6 weeks.
  Interventions: Device: I-BiTTM DVD

INTERVENTIONS:
Device: I-BiTTM game — 30 minutes intervention weekly for 6 weeks.
  Arms: I-BiTTM game
Device: Non-I-BiTTM game — 30 minutes intervention weekly for 6 weeks.
  Arms: Non-I-BiTTM game
Device: I-BiTTM DVD — 30 minutes intervention weekly for 6 weeks.
  Arms: I-BiTTM DVD

SUMMARY:
The study aims to determine whether 30 minutes of treatment playing an interactive computer game weekly for 6 weeks, improves visual acuity. The game has been specially configured to ensure the amblyopic eye is preferentially stimulated and the patient wears shutter glasses which manipulate the image seen by each eye in order to provide more information to the amblyopic eye. Patients will be randomised to play the computer game using the I-BiTTM technology, play the computer game but without the I-BiTTM technology, or watch a DVD using the I-BiTTM technology.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of Anisometropic, Strabismic or Mixed Amblyopia as made by an Orthoptist
* Male or Female
* Aged 4 - 8 years inclusive.
* Participant's parent or guardian is willing and able to give informed consent for participation in the study

Exclusion criteria:

* Stimulus deprivation amblyopia.
* Organic lesions of the eye preventing the establishment of good vision (e.g. media opacities, abnormalities in the fundus or optic nerve).
* Lesions of the brain preventing the establishment of good vision (e.g. cortical visual impairment).
* Patients diagnosed with Photosensitive Epilepsy
* Patients diagnosed with or suspected of having Conjunctivitis
* Loss of suppression at filter 4 or less as measured with the Sbisa Bar
* Establishment of normal vision by refractive adaptation (wearing glasses after presentation).
* Inability to comply with the follow up visits required
* Refusal to accept randomisation
* Have participated in a previous study examining I-BiT treatment

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual acuity | 6 weeks

SECONDARY OUTCOMES:
Change from baseline in visual acuity | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Foss, BA BMBCh MRCP MRCOphth FRC, Principal Investigator — Consultant Ophthalmologist
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Trust, Cambridge, Cambridgeshire
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire

REFERENCES:
- [Derived] Tailor V, Ludden S, Bossi M, Bunce C, Greenwood JA, Dahlmann-Noor A. Binocular versus standard occlusion or blurring treatment for unilateral amblyopia in children aged three to eight years. Cochrane Database Syst Rev. 2022 Feb 7;2(2):CD011347. doi: 10.1002/14651858.CD011347.pub3. PMID 35129211
- [Derived] Herbison N, MacKeith D, Vivian A, Purdy J, Fakis A, Ash IM, Cobb SV, Eastgate RM, Haworth SM, Gregson RM, Foss AJ. Randomised controlled trial of video clips and interactive games to improve vision in children with amblyopia using the I-BiT system. Br J Ophthalmol. 2016 Nov;100(11):1511-1516. doi: 10.1136/bjophthalmol-2015-307798. Epub 2016 Mar 7. PMID 26951772
- [Derived] Foss AJ, Gregson RM, MacKeith D, Herbison N, Ash IM, Cobb SV, Eastgate RM, Hepburn T, Vivian A, Moore D, Haworth SM; I-BiT Steering group. Evaluation and development of a novel binocular treatment (I-BiT) system using video clips and interactive games to improve vision in children with amblyopia ('lazy eye'): study protocol for a randomised controlled trial. Trials. 2013 May 20;14:145. doi: 10.1186/1745-6215-14-145. PMID 23688108
- See also: Project website — http://www.lazy-i-bit.com/